CLINICAL TRIAL: NCT07181746
Title: Effect of Pilates Exercises on Restless Leg Syndrome, Functional Capacity and Physical Self-perception Among Older Adult Undergoing Hemodialysis
Brief Title: Effect of Exercises on Restless Leg Syndrome, Functional Capacity and Physical Self-perception Among Hemodialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norther Private Collage of Nursing (Other)
Responsible Party: Principal Investigator, Amal Hashem, Associate professor, Norther Private Collage of Nursing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: amalhasem@nec.edu.sa
Record Dates: First submitted 2025-09-06; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Hemodialysis; Functional Capacities; Excercise

STUDY DESIGN:
Intervention Model Description: single group assignment
Masking Description: Non
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Active Comparator): Pilates Exercises
  Interventions: Procedure: leg exercises

INTERVENTIONS:
Procedure: leg exercises — The patient in study group will offer 72 planned sessions along 16-week period, each session consisted of 5 minutes walking as a warm-up, followed by 30 to 45 minutes of resistance exercises tolerated by the patient, time maintained until the end of the intervention. Each participant will receive about two to three, personal training session regarding the technique of resistance training until they are perfect in performing the exercises. Participants will receive a booklet with instructions on the Pilates training illustrated by colored pictures. The sessions during the staying the patient's in the hospital will be supervised by the researchers

SUMMARY:
The study aimed to evaluate the effect of Pilates exercises on restless leg syndrome, functional capacity and physical self-perception among older adult undergoing hemodialysis. participants are 60 elderly patients both male and female who undergoing maintenance hemodialysis.

DETAILED DESCRIPTION:
The research hypothesis include : H1: Older Adult Undergoing Hemodialysis who will practice Pilates exercises will have less severity of the Restless Leg Syndrome, and high Functional Capacity and Physical Self-Perception than those who will not practice.

Participants were divided into two groups (study and control). Both groups were asked to fill out all questionnaires before and after the study using the same tools. In the control group, older adult receives routine care, which was provided by the hospital as examination, routine medication . Participants were asked to answer a post-test using the same pre-test questionnaires. And the study group were divided into small training groups with 3-5 older adult for each group.

ELIGIBILITY:
Inclusion Criteria:

* • Age of ≥ 65 years old,

  * A History of hemodialysis treatment two to three times per week for at least six months,
  * Interest in participation,
  * Being able to move independently and with a physical condition certified by a physician to play the sport, with no myocardial infarction or surgery in the past six months of the study.

Exclusion Criteria:

* Three or more absences in exercise sessions;
* Being a habitual Pilates practitioner;
* Detection of reduced exercise tolerance, including tachycardia, shortness of breath, and feeling too tired or weak;
* Peritoneal dialysis during the study; and other concurrent clinical conditions, such as cardio-respiratory problems reported by physician and/or patients

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-02 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
change in severity level of restless leg syndrome | 3 month
  Restless Leg Syndrome Rating Scale: used for assessing the severity restless legs syndrome (RLS). This tool composed of 10-item questionnaire asks respondents to use Likert-type ratings. Each question contains answers that score from 0 to 4 points, with 0 representing the absence of a problem and 4 representing a very severe problem. Total scores can range from 0 to 40. Questions can be divided into one of two categories: disorder symptoms (nature, intensity, and frequency) and their impact (sleep issues, disturbances in daily functioning, and resultant changes in mood). Very severe=31-40 points, Severe=21-30 points, Moderate=11-20 points, Mild=1-10 points, None=0 points

IPD SHARING:
Plan to Share IPD: No